CLINICAL TRIAL: NCT01008267
Title: Shockwave Lithotripsy (SWL) Under Regular General Anesthesia and Under General Anesthesia Using Bronchial Blocker.
Brief Title: Shockwave Lithotripsy (SWL) Under Selective, General Anesthesia.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Zoya Haitov MD, Anesthesiology department, Assaf-Harofeh Medical Center
Other Study IDs: 63/09
Record Dates: First submitted 2009-11-04; First posted 2009-11-05 (Estimated); Last update posted 2009-11-05 (Estimated); Status verified 2009-03

CONDITIONS: Renal Calculi; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- SWL under general anesthesia: Patients who failed in SWL under sedation(a standard protocol), will undergo a second SWL process under general anesthesia.
- SWL under general selective anesthesia: Patients who failed in SWL under sedation(a standard protocol), will undergo a second SWL process under general selective anesthesia, using a bronchial blocker.

SUMMARY:
SWL is widely used in the treatment of patients with renal and ureteral calculi. Several factors determine the success of extracorporeal shockwave lithotripsy (SWL) for kidney stones: stone size, stone location within the collecting system, stone type, and the SWL machine used. Moreover, in some cases it is very difficult to focus on the stone because of its movement as a results of breathing. In order to prevent stone movement we want to use a bronchial blocker, processing a selective ventilation of the opposite side of stone location.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Not pregnant
* All patients who failed in SWL process, taken under sedation (standard protocol)

Exclusion Criteria:

* Age < 18
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who failed in SWL process taken under sedation (standard protocol)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology department, Assaf-Harofeh MC, Beer-Yaakov, Zrifin, Israel